CLINICAL TRIAL: NCT05573607
Title: Effects of a Dietary Supplement Containing Salacia Extract, Citrus Bioflavonoids, and Trivalent Chromium on Markers of Glucose Control and Quality of Life: A Randomized, Placebo-Controlled, Double-Blind Pilot Study
Brief Title: Effects of a Dietary Supplement on Markers of Glucose Control and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Collaborators: Mend Nutrition, Inc (Unknown); Keller Consulting Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 25-CAHS-104
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Blood Glucose
MeSH Terms: interventions — Chromium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Consists of a maltodextrin tablet
  Interventions: Dietary Supplement: Placebo
- Active (Active Comparator): A tablet consisting of a blend of Crominex® 3+, Capros® Amla Extract (Fruit), PrimaVie® Shilajit), and MetaviveTM complex (Salacia Chinensis Extract (Fruit) and a Citrus Bioflavonoids)
  Interventions: Dietary Supplement: Chromium

INTERVENTIONS:
Dietary Supplement: Placebo — Maltodextrin tablet
  Arms: Placebo
Dietary Supplement: Chromium — A tablet consisting of a blend of Crominex® 3+, Capros® Amla Extract (Fruit), PrimaVie® Shilajit), and MetaviveTM complex (Salacia Chinensis Extract (Fruit) and a Citrus Bioflavonoids)
  Arms: Active

SUMMARY:
This study is a double-blind, randomized, two-arm, placebo-controlled trial of apparently healthy men and women to be recruited at a single investigational center in Northeast Ohio (i.e. The Center for Applied Health Sciences). Subjects will attend four study visits. During Visit 1, subjects will be screened for participation (i.e., medical history, physical exam, routine blood work [also HgA1c, insulin], background baseline diet). Over the next 12 weeks, subjects will attend Visits 2-4, wherein assessments of serum glucose, insulin, HOMA-IR, 2-hour glucose tolerance test (GTT), HgA1c, C-reactive protein, adiponectin, ferritin, waist circumference, quality of life questionnaire, and various visual analog scales for appetite, satiety, and cravings will be made.

ELIGIBILITY:
Inclusion Criteria:

Provide voluntary signed and dated informed consent. Be in good health as determined by medical history and routine blood chemistries.

Age between the ages of 21 and 65 (inclusive). Body Mass Index of 18.5-34.99 (inclusive). Body weight of at least 120 pounds. Fasting blood sugar of 100-125 (inclusive) OR HgA1c of 5.7-6.4% (inclusive). Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic bloodpressure < 90 mm Hg.

Normal seated, resting heart rate (<90 per minute). Willing to duplicate their previous 24-hour diet, refrain from caffeine for 12 hrs and exercise for 24 hr prior to each trial, and fast for 10 hours prior each of the treatments.

Exclusion Criteria:

History of unstable or new-onset cardiovascular or cardiorespiratory disease. History of diabetes, or other endocrine disorder. Fasting blood sugar of > 125 mg/dL or HgA1c of > 6.4%. History of use of medications or dietary supplements known to affect glycemia or insulinemia.

History of hyperparathyroidism or an untreated thyroid disease. History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).

Prior gastrointestinal bypass surgery (Lapband), etc. Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g. short bowel syndrome, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).

Chronic inflammatory condition or disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).

Known sensitivity to any ingredient in the test formulations as listed in the Certificates-of- Analysis.

Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.

Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
glucose | change from baseline to week 12
  measurement of glucose in blood
insulin | change from baseline to week 12
  measurement of insulin in blood

SECONDARY OUTCOMES:
cravings | change from baseline to week 12
  cravings as measured with a 10 cm anchored visual analogue scale, where higher values represent greater cravings.
satiety | change from baseline to week 12
  satiety as measured with a 10 cm anchored visual analogue scale, where higher values represent greater cravings.
adiponectin | change from baseline to week 12
  measurement of adiponectin in blood
blood urea nitrogen | change from baseline to week 12
  measurement of blood urea nitrogen in blood
creatinine | change from baseline to week 12
  measurement of creatinine in blood
alanine aminotransferase | change from baseline to week 12
  measurement of alanine aminotransferase in blood
aspartate aminotransferase | change from baseline to week 12
  measurement of aspartate aminotransferase in blood
Short Form Health Survey (SF-36) | change from baseline to week 12
  health status as measured with the SF-36 questionnaire, where scores range from 0 to 100, and higher values represent better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided